CLINICAL TRIAL: NCT01520376
Title: A Prospective Randomized Trial to Asses the Efficacy of an Early Psychiatric Counseling Compared to Usual Care in a Cohort of Patients Hospitalized for an Acute Exacerbation of COPD in Prevention of Re-exacerbation
Brief Title: Anxiety and Depression in Patients Hospitalizes for an Acute Exacerbation of COPD
Acronym: ADPHA-EPOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nestor Soler Porcar, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Nestor Soler Porcar, MD, PhD, Especialista Sènior, Fundacion Clinic per a la Recerca Biomédica
Organization: Fundacion Clinic per a la Recerca Biomédica (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ADPHA-EPOC
Record Dates: First submitted 2012-01-25; First posted 2012-01-27 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Chronic Obstructive Pulmonary Disease; Anxiety; Depression
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Anxiety Disorders; Depression | interventions — Counseling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Counselling (Active Comparator): People receiving a psychiatric evaluation after screening (HADS test > 12 points) and revised at 1 and 6 months
  Interventions: Behavioral: Counselling
- Usual care (No Intervention): People after screening (HADS test > 12 points) and send to their primary care physician

INTERVENTIONS:
Behavioral: Counselling — Visit by a psychiatrist at day-30 and day-180 after discarge
  Arms: Counselling

SUMMARY:
This study will try to elucidate wheter the impact of a psychiatric intervention in patients hospitalized because an acute exacerbation of COPD and anxiety/depression and reconsulting at 1 and 6 month after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of any ethnic group
* Above 40 years old
* Diagnose with Chronic Obstructive Pulmonary disease (COPD) according to the ATS/ERS guidelines
* Acute exacerbation of COPD according to the following criteria:

  a) Cyanosis b) Obnubilations or mental confusion d) Respiratory Rate above 25 per minute e) Failure of ambulatory treatment f) Co-morbidities that worsens respiratory condition g) Dyspnea

Exclusion Criteria:

* Less than 6 months expectancy of life
* Needing of mechanical ventilation
* Severe cardiovascular disease
* Pregnancy
* Previous diagnosis of depression/anxiety

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2011-10; Primary Completion 2013-10 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Efficacy of the intervention | 6 months
  Counselling vs. usual care on re-hospitalizations

SECONDARY OUTCOMES:
Impact of diagnosis | 6 months
  Anxiety/depression diagnosis on number of exacerbations at 1 and 6 months, comparing patients with screening on HADS test > 12

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Huerta, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Fundacio Clinic Per la Recerca Biomèdica - Hospital Clinic de Barcelona, Barcelona, Catalonia, Spain